CLINICAL TRIAL: NCT03124225
Title: The Impact of Rheumatologist-performed Ultrasound on Diagnosis and Management of Inflammatory Arthritis in Routine Clinical Practice
Brief Title: Ultrasound Utility in Routine Clinical Practise
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IMM 09-0270
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2016-09

CONDITIONS: Arthritis, Rheumatoid; Ultrasonography
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ultrasound: Early Arthritis Patients seeing a Rheumatologist who uses US for assessment routinely in clinic
  Interventions: Drug: DMARD
- Non-Ultrasound: Early Arthritis Patients seeing a Rheumatologist who does not uses US for assessment routinely in clinic
  Interventions: Drug: DMARD

INTERVENTIONS:
Drug: DMARD

SUMMARY:
The aim of this research study is to describe the impact of rheumatologist performed ultrasound on the diagnosis and management pathways of patients with rheumatoid arthritis. Primarily, to compare the time from first visit to treatment initiation between patients with and without rheumatologist-performed ultrasound assessment.

DETAILED DESCRIPTION:
There are currently no guidelines for best practice in the use of ultrasound in RA and interim results from a survey by the British Society of Rheumatology (BSR) in this area have suggested that practice is variable across the UK. NICE recognize that the earlier persistent synovitis is identified and treated with disease modifying anti-rheumatic drugs DMARDs, the better the long term outcome and have welcomed the need to determine the role of imaging in assisting with this early diagnosis, and whether the added cost is justified by better disease outcomes.

This is a multi-site prospective observational study which investigates the use of ultrasound imaging in the context of patients with early arthritis presenting to secondary care. The time to commencement of DMARD therapy and diagnosis of Rheumatoid arthritis are therein outcome measures. Patients are followed up for 12 months after their first presentation and time to diagnosis or DMARD commencement recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years at the time of presentation to the clinic Patients newly presenting to the rheumatology clinic with suspected inflammatory arthritis

Exclusion Criteria:

* For the non-ultrasound arm; patients who have been referred to another rheumatologist or radiologist for ultrasound Patients who decline or who are unable to consent to the use of their medical records for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early Arthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To compare the time from first visit to treatment initiation between patients with and without rheumatologist-performed ultrasound assessment | 12 months